CLINICAL TRIAL: NCT03750552
Title: A Phase 3, 4-week, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study of TD-9855 in Treating Symptomatic Neurogenic Orthostatic Hypotension in Subjects With Primary Autonomic Failure
Brief Title: Clinical Effect of Ampreloxetine (TD-9855) for Treating Symptomatic nOH in Subjects With Primary Autonomic Failure
Acronym: SEQUOIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0169; 2018-003289-15 (EudraCT Number)
Record Dates: First submitted 2018-11-20; First posted 2018-11-23 (Actual); Results first posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-08

CONDITIONS: Symptomatic Neurogenic Orthostatic Hypotension
Keywords: Symptomatic Neurogenic Orthostatic Hypotension; symptomatic nOH; multiple system atrophy; MSA; Parkinson's disease; PD; pure autonomic failure; PAF; primary autonomic failure; SEQUOIA; ampreloxetine; low blood pressure; dizziness; fainting; blacking out; lightheadedness; norepinephrine; hypotension; Parkinsonism; TD-9855; Neurogenic Orthostatic Hypotension; nOH; 0145; 145; 169; 0169; TD9855
MeSH Terms: conditions — Multiple System Atrophy; Parkinson Disease; Pure Autonomic Failure; Hypotension; Dizziness; Syncope; Parkinsonian Disorders | interventions — ampreloxetine

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ampreloxetine (Experimental): Participants randomized to ampreloxetine will receive a single, oral, daily dose of active drug for 4 weeks.
  Interventions: Drug: ampreloxetine
- Placebo (Placebo Comparator): Participants randomized to Placebo will receive a single, oral, daily dose of placebo for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ampreloxetine — Oral tablet, QD
  Other Names: TD-9855
  Arms: ampreloxetine
Drug: Placebo — Oral tablet, QD
  Arms: Placebo

SUMMARY:
A Phase 3 study to evaluate efficacy, safety, and tolerability of ampreloxetine (TD-9855) in subjects with primary autonomic failures (MSA, PD, or PAF) and symptomatic nOH with up to 4 weeks of treatment.

DETAILED DESCRIPTION:
A Phase 3, randomized, double-blind, placebo-controlled, parallel-group, multicenter study to evaluate efficacy, safety, and tolerability of ampreloxetine (TD-9855) in subjects with primary autonomic failures (MSA, PD, or PAF) and symptomatic nOH. The study consists of 3 periods: (i) 4-week screening, (ii) 4-week randomized treatment, and (iii) 2-week follow up. The trial utilizes an operational design featuring the ability to conduct protocol required visits as either in clinic or remote visits (except Screening visit).

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female and at least 30 years old.
* Subject must meet the diagnostic criteria of symptomatic nOH, as demonstrated by a sustained reduction in BP of ≥20 mm Hg (systolic) or ≥10 mm Hg (diastolic) within 3 minutes of being tilted-up to ≥60o from a supine position as determined by a tilt-table test.
* Subject must score at least a 4 on the Orthostatic Hypotension Symptom Assessment Question #1 at randomization visit.
* For subjects with PD only: Subject has a diagnosis of PD according to the United Kingdom Parkinson's Disease Society (UKPDS) Brain Bank Criteria (1992).
* For subjects with MSA only: Subject has a diagnosis of possible or probable MSA of the Parkinsonian subtype (MSA-P) or cerebellar subtype (MSA-C) according to The Gilman Criteria (2008).
* For subjects with PAF only: Subject has documented impaired autonomic reflexes, including the Valsalva maneuver performed within 24 months from the date of randomization.
* Subject has plasma NE levels >100 pg/mL after being in seated position for 30 minutes.

Exclusion Criteria:

* Subject has a known systemic illness known to produce autonomic neuropathy, including but not limited to amyloidosis, and autoimmune neuropathies.
* Subject has a known intolerance to other NRIs or SNRIs.
* Subject currently uses concomitant antihypertensive medication for the treatment of essential hypertension unrelated to autonomic dysfunction.
* Subject has used strong CYP1A2 inhibitors or inducers within 7 days or 5 half-lives, whichever is longer, prior to randomization or requires concomitant use until the follow-up visit.
* Subject has changed dose, frequency, or type of prescribed medication for orthostatic hypotension within 7 days prior to V1.

  * Midodrine and droxidopa (if applicable) must be tapered off at least 7 days prior to V1.
* Subject has a known or suspected alcohol or substance abuse within the past 12 months (DSM-IV-TR® definition of alcohol or substance abuse).
* Subject has a clinically unstable coronary artery disease, or major cardiovascular or neurological event in the past 6 months.
* Subject has used any monoamine oxidase inhibitor (MAO-I) within 14 days prior to randomization.
* Subject has a history of untreated closed angle glaucoma, or treated closed angle glaucoma that, in the opinion of an ophthalmologist, might result in an increased risk to the subject.
* Subject has any significant uncontrolled cardiac arrhythmia.
* Subject has a Montreal Cognitive Assessment (MoCA) ≤23.
* Subject had a myocardial infarction in the past 6 months or has current unstable angina.
* Subject has known congestive heart failure (New York Heart Association [NYHA] Class 3 or 4).
* Subject has a clinically significant abnormal laboratory findings (e.g., alanine aminotransferase [ALT] or aspartate aminotransferase [AST] >3.0 x upper limit of normal [ULN]; blood bilirubin [total] >1.5 x ULN; estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m2, or any abnormal laboratory value that could interfere with safety of the subject).
* Subject has demonstrated a history of lifetime suicidal ideation and/or suicidal behavior, as outlined by the C-SSRS (Columbia Suicide Severity Rating Scale) (Baseline/Screening Version) subject should be assessed by the rater for risk of suicide and the subject's appropriateness for inclusion in the study.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (125):
- United States (23):
  - Banner Sun Health Research Institute, Sun City, Arizona
  - Collaborative Neuroscience Network, LLC, Long Beach, California
  - Stanford Neuroscience Health Center, Palo Alto, California
  - Colorado Springs Neurological Associates, PC, Colorado Springs, Colorado
  - University of Colorado Health, Loveland, Colorado
  - Georgetown University Hospital, Dept. of Neurology, Washington D.C., District of Columbia
  - Parkinson's Disease and Movement Disorders Center, Boca Raton, Florida
  - SFM Clinical Research, Boca Raton, Florida
  - Fixel Institute for Neurological Diseases, Gainesville, Florida
  - Neurostudies, Inc, Port Charlotte, Florida
  - Rush University Medical Center, Chicago, Illinois
  - NorthShore University Health System, Glenview, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - New York University Langone Health, New York, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Georgetown University Hospital, McLean, Virginia
  - Inland Northwest Research, Spokane, Washington
- Australia (5):
  - Concord Hospital, Concord, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Monash Health - Clinical Trials Centre, Clayton, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
  - Perron Institute for Neurological and Translational Science, QEII Medical Centre, Nedlands
- Austria (3):
  - Medizinische Universitat Innsbruck Abteilung Fur Neurologie, Innsbruck
  - Universitätsklinikum Tulln, Tulln
  - Wilhelminenspital Wien Abteilung fur Neurologie, Vienna
- Bulgaria (3):
  - UMHAT Sveti Georgi EAD Clinic of Neurological Diseases, Plovdiv
  - MHATNP Sv.Naum, EAD, Sofia
  - UMHAT Alexandrovska EAD Clinic of Neurological Diseases, Sofia
- Canada (4):
  - University of Calgary, Calgary, Alberta
  - London Health Sciences Centre-CCIT, London, Ontario
  - University Health Network - Toronto Western Hospital Movement Disorders Clinic, Toronto, Ontario
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
- Denmark (2):
  - Bispebjerg og Frederiksberg Hospital, Copenhagen
  - Odense Universitetshospital, Odense
- Estonia (3):
  - East Tallinn Central Hospital, Tallinn
  - Astra Team Clinic, Tallinn
  - Tartu University Hospital, Tartu
- France (3):
  - Hopital Roger Salengro - CHU Lille, Lille, Nord
  - CHU Caremeau, Nîmes
  - Hospital Pierre Paul Rquet, CHU Purpan, Toulouse
- Germany (7):
  - Universitaetsklinikum Freiburg - Klinik fur Neurologie und Neurophysiologie, Freiburg im Breisgau, Baden-Wurttemberg
  - Gemeinschaftspraxis Dr. med. J. Springub/ W. Schwarz, Westerstede, Lower Saxony
  - Praxis Dr. Oehlwein, Gera, Thuringia
  - Charite Universitatsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - Alexianer St. Joseph-Krankenhaus Berlin-Weißensee, Klinik für Neurologie, Berlin
  - Charite - Campus Virchow-Klinikum, Klinik fur Neurologie, Berlin
  - Charite - Campus Virchow-Klinikum, Berlin
- Hungary (4):
  - Clinexpert Kft., Budapest
  - Semmelweis Egyetem, Budapest
  - Pecsi Tudomanyegyetem, Neurologiai Klinika, Pécs
  - Szent Borbala Korhaz, Tatabánya
- Israel (5):
  - Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Ziv Medical Center, Safed
  - Tel Aviv Medical Center, Tel Aviv
  - Chaim Sheba Medical Center, Tel Litwinsky
- Italy (17):
  - Istituto Clinico Humanitas - IRCCS, Rozzano, Milano
  - Fondazione Istituto G.Giglio di Cefalù, Cefalù, Palermo
  - Azienda Ospedaliero Universitaria Ospedali Riuniti Ancona Umberto I - G.M. Lancisi - G. Salesi, SOD Clinica di Neuroriabilitazione, Ancona
  - Universita di Bologna-Clinica Neurologica-Dipartimento di Scienze Neurologiche Ospedale Bellaria, Bologna
  - Azienda Ospedaliero - Universitaria Policlinico Vittorio Emanuele. - P.O G. Rodolico, Clinica Neurologica, Catania
  - Universita Gabriele D'Annunzio- Cesi-Met, Chieti
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale San Raffaele I U.O. di Neurologia, Milan
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Fondazione PTV - Policlinico Tor Vergata I U.O.C. Neurologia, Roma
  - Ospedale San Giovanni Battista del Sovrano Militare Ordine di Malta, Roma
  - Ospedale San Giovanni Battista, Roma
  - Policlinico Umberto I - Universita degli Studi di Roma La Sapienza / Neurologia, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS / Istituto di Neurologia - Ambulatorio Disturbi del Movimento, Roma
  - Sapienza University of Rome, Roma
  - AOU San Giovanni di Dio e Ruggi d'Aragona, Salerno
  - A.O. Santa Maria, Terni
- New Zealand Brain Research Institute, Christchurch, New Zealand
- Poland (8):
  - Specjalistyczna Praktyka Lekarska prof.Grzegorz Opala, Katowice
  - PRATIA MCM Kraków, Krakow
  - Krakowska Akademia Neurologii Sp z o.o. Centrum Neurologii Klinicznej, Krakow
  - Samodzielny Publiczny Szpital Kliniczny Nr 4 w Lublinie, Lublin
  - Instytut Zdrowia dr Boczarska-Jedynak, Oświęcim
  - NEURO-CARE Sp. z o.o. Sp. Komandytowa, Siemianowice Śląskie
  - ETG Warszawa, Warsaw
  - Specjalistyczne Gabinety sp. z o.o., Warsaw
- Portugal (3):
  - Hospital Senhora da Oliveira - Guimaraes, EPE, Guimarães
  - Centro Hospitalar e Universitario Lisboa Norte - Hospital de Santa Maria, Lisbon
  - Campus Neurologico Senior, Torres Vedras
- Russia (10):
  - State Autonomous Institution of Healthcare Republican Clinical Hospital of the Ministry of Healthcare of Republic Tatarstan, Kazan', Tatarstan Republic
  - Federal State Budgetary Institution Federal Sibirian Scientific and Clinical Center of Federal Medico-Biological Agency, Krasnoyarsk
  - Federal State Budgetary Educational Institution of Additional Professional Education Russian Medical Academy of Continuous Postgraduate Education of the Ministry of Healthcare of the Russian Federation, Moscow
  - NHI Central Clinical Hospital #2 of JSC Russian Railways N.A. Semashko, Moscow
  - City Neurological Center Sibneiromed, Novosibirsk
  - SBEIHPE Novosibirsk State Medical University, Novosibirsk
  - Federal State Budgetary Institution National Medical Research Centre of psychiatry and neurology named after V.M. Bekhterev of the Ministry of Healthcare of the Russian Federation, Saint Petersburg
  - Human Brain Institute RAMS, Saint Petersburg
  - Saint Petersburg State Budgetary Institution of Healthcare City Hospital # 40 of Kurortnyi Region, Saint Petersburg
  - Regional State Budgetary Institution of Healthcare Smolensk Regional Clinical Hospital, Smolensk
- Spain (11):
  - Hospital Universitario Donostia, San Sebastián, Guipuzcoa
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Navarrabiomed Fundacion Miguel Servet, Pamplona, Navarre
  - Hospital de Cruces, Barakaldo, Vizcaya
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Mutua de Terrasa, Barcelona
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital Universitario de La Princesa, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
- Ukraine (5):
  - Communal Institution Dnipropetrovsk I.I.Mechnikov RCH, Dnipro
  - Communal Noncommercial Enterprise City Policlinic #9 of Kharkiv City Council, Kharkiv
  - Communal Noncommercial Enterprise of Lviv Regional Council Lviv Regional Clinical Hospital Dept of Neurology, Lviv
  - CNE Acad O.I. Yushchenko Vinnytsia Reg Psychoneurological Hospital of Vinnytsia Regional Council, Department of Neurology, Vinnytsia
  - Communal Institution City Clinical Hospital #6, Zaporizhzhia
- United Kingdom (8):
  - Royal Devon and Exeter Hospital, Exeter, Devon
  - Re:Cognition Health, Plymouth, Devon
  - Barts Hospital, London, Greater London
  - The National Hospital for Neurology & Neurosurgery, London, Greater London
  - King's College Hospital, London, Manchester
  - Re:Cognition Health Ltd, Birmingham, West Midlands
  - Re:Cognition Health, London
  - Salford Royal, Salford

IPD SHARING:
Plan to Share IPD: No
Theravance Biopharma, Inc. will not be sharing individual de-identified participant data or other relevant study documents.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 195 participants were enrolled across 76 sites in Australia, Austria, Bulgaria, Canada, Denmark, Estonia, France, Germany, Hungary, Israel, Italy, New Zealand, Poland, Portugal, Spain, Russia, Ukraine, United Kingdom and the United States.
Pre-assignment Details: Overall, 194 randomized participants received at least one dose of study drug. Eight participants from one site were excluded from all analysis sets except the Randomized Analysis Set due to data integrity concerns.
Groups:
- Ampreloxetine: Participants received ampreloxetine at a dose of 10 mg once daily (QD) for 4 weeks.
  Ampreloxetine: Oral tablet, QD
- Placebo: Participants received placebo QD for 4 weeks. Placebo: Oral tablet, QD
Period: Overall Study
Arm/Group | Ampreloxetine | Placebo
Started | 98 | 97
Safety Analysis Set | 96 | 90
Full Analysis Set | 94 | 90
Completed | 90 | 95
Not Completed | 8 | 2
Not completed — Adverse Event | 5 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Other | 2 | 0

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population includes all participants from the Randomized Analysis Set.
Groups:
- Placebo: Participants received placebo once daily (QD) for 4 weeks. Placebo: Oral tablet, QD
- Total: Total of all reporting groups
Arm/Group | Ampreloxetine | Placebo | Total
Number analyzed (Participants) | 98 | 97 | 195
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 28 | 25 | 53
  ≥ 65 years | 70 | 72 | 142
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 29 | 66
  Male | 61 | 68 | 129
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 92 | 91 | 183
  Unknown or Not Reported | 5 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 96 | 94 | 190
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Orthostatic Hypotension Symptom Assessment (OHSA) Question #1 Score at Week 4
Description: OHSA is an assessment of the severity of symptoms from low blood pressure. OHSA is a 6 question symptom assessment scale where each question uses an 11 point scale from 0 to 10, with 0 indicating no symptoms/no interference and 10 indicating the worst possible symptoms/complete interference.
  Question #1 assesses dizziness, lightheadedness, feeling faint, or feeling like you might blackout.
  A mean negative change from baseline indicates a better outcome.
Time Frame: Baseline and Week 4
Population: Participants included in the Full Analysis Set, defined as all randomized participants who received at least one dose of study medication and had at least 1 post-baseline measurement of Orthostatic Hypotension Symptom Assessment (OHSA) question 1, were included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Ampreloxetine | Placebo
Number analyzed (Participants) | 94 | 90
score on a scale | -1.69 (0.290) | -1.45 (0.293)
Statistical Analysis 1: Comparison: Ampreloxetine vs Placebo; Test type: Superiority; p = 0.574, Mixed Model Repeated Measures; Least Squares Mean Difference = -0.23, 95% CI 2-sided [-1.05 to 0.58], Standard Error of Mean 0.413

2. Secondary Outcome: Change From Baseline in Orthostatic Hypotension Symptom Assessment (OHSA) Composite Score at Week 4
Description: OHSA is an assessment of the severity of symptoms from low blood pressure. OHSA is a 6 question symptom assessment scale in which the composite score uses an 11 point scale from 0 to 10, with 0 indicating no symptoms/no interference and 10 indicating the worst possible symptoms/complete interference.
  A mean negative change from baseline indicates a better outcome.
Time Frame: Baseline and Week 4
Population: Participants included in the Full Analysis Set, defined as all randomized participants who received at least one dose of study medication and had at least 1 post-baseline measurement of Orthostatic Hypotension Symptom Assessment (OHSA) question 1, with a valid composite OHSA score at Week 4 were included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Ampreloxetine | Placebo
Number analyzed (Participants) | 90 | 87
score on a scale | -1.32 (0.200) | -1.05 (0.202)
Statistical Analysis 1: Comparison: Ampreloxetine vs Placebo; Test type: Superiority; p = 0.331, Mixed Model Repeated Measures; Least Squares Mean Difference = -0.28, 95% CI 2-sided [-0.84 to 0.28], Standard Error of Mean 0.284

3. Secondary Outcome: Change From Baseline in Orthostatic Hypotension Daily Activities Scale (OHDAS) Composite Score at Week 4
Description: OHDAS is an assessment of how low blood pressure symptoms affect daily life. OHDAS is a 4 item assessment in which the composite score uses an 11 point scale from 0 to 10, with 0 indicating no symptoms/no interference and 10 indicating the worst possible symptoms/complete interference.
  A mean negative change from baseline indicates a better outcome.
Time Frame: Baseline and Week 4
Population: Participants included in the Full Analysis Set, defined as all randomized participants who received at least one dose of study medication and had at least 1 post-baseline measurement of Orthostatic Hypotension Symptom Assessment (OHSA) question 1, with a valid composite OHDAS score at Week 4 were included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Ampreloxetine | Placebo
Number analyzed (Participants) | 87 | 85
score on a scale | -1.22 (0.265) | -0.95 (0.267)
Statistical Analysis 1: Comparison: Ampreloxetine vs Placebo; Test type: Superiority; p = 0.481, Mixed Model Repeated Measures; Least Squares Mean Difference = -0.27, 95% CI 2-sided [-1.01 to 0.48], Standard Error of Mean 0.376

4. Secondary Outcome: Number of Participants Who Experienced an Improvement From Baseline in Patient Global Impression of Change (PGI-C) Score at Week 4
Description: PGI-C was assessed using a 5-point scale where participants were asked to compare their current condition to their condition at baseline from 1 to 5, with 1 indicating the condition is very much improved and 5 indicating the condition is very much worse. These scores were analyzed in 2 categories: better and no change/worse.
Time Frame: Baseline and Week 4
Population: Participants included in the Full Analysis Set, defined as all randomized participants who received at least one dose of study medication and had at least 1 post-baseline measurement of Orthostatic Hypotension Symptom Assessment (OHSA) question 1, who have available data were included in this analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Participants receives placebo once daily (QD) for 4 weeks. Placebo: Oral tablet, QD
Arm/Group | Ampreloxetine | Placebo
Number analyzed (Participants) | 91 | 87
Participants | 49 | 45
Statistical Analysis 1: Comparison: Ampreloxetine vs Placebo; Test type: Superiority; p = 0.740, Cochran-Mantel-Haenszel; Stratified by disease type; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.12 to 0.17], Standard Error of Mean 0.073 — The assumed common risk difference estimate and standard error are calculated using Mantel-Haenszel stratum weights and the Sato variance estimator. Mantel-Haenszel confidence limits are shown

5. Secondary Outcome: Number of Participants Who Experienced at Least One Fall
Time Frame: Up to Week 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Ampreloxetine | Placebo
Number analyzed (Participants) | 93 | 90
Participants | 33 | 22
Statistical Analysis 1: Comparison: Ampreloxetine vs Placebo; Test type: Superiority; p = 0.0903, Cochran-Mantel-Haenszel; Stratified by disease type; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.02 to 0.24], Standard Error of Mean 0.064 — [estimate comment as in outcome 4, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to Day 43
Description: Participants in the Safety Analysis set, defined as all randomized subjects who received at least 1 dose of study medication, were included in this analysis.
Arm/Group | Ampreloxetine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/96 | 0/90
Serious Adverse Events (participants affected / at risk) | 4/96 | 2/90
Other Adverse Events (participants affected / at risk) | 42/96 | 38/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ampreloxetine (N=96) | Placebo (N=90)
Pneumonia (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Asthenia (General disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ampreloxetine (N=96) | Placebo (N=90)
Headache (Nervous system disorders) | 5 | 3
Urinary tract infection (Infections and infestations) | 3 | 4
Fatigue (General disorders) | 3 | 1
Insomnia (Psychiatric disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 2 | 2
Supine hypertension (Vascular disorders) | 1 | 3
Anxiety (Psychiatric disorders) | 2 | 1
Asthenia (General disorders) | 1 | 1
Dizziness (Nervous system disorders) | 3 | 0
Hypertension (Vascular disorders) | 3 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Blood creatinine phosphokinase increased (Investigations) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Somnolence (Nervous system disorders) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abnormal dreams (Psychiatric disorders) | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0
Bacterial disease carrier (Infections and infestations) | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 1
Bladder pain (Renal and urinary disorders) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
Blood urea increased (Investigations) | 0 | 1
Blood urea nitrogen/creatine ratio increased (Investigations) | 1 | 0
Bulbar palsy (Nervous system disorders) | 1 | 0
Catheter site pain (General disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Crystal urine present (Investigations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Disorientation (Psychiatric disorders) | 0 | 1
Dizziness postural (Nervous system disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Eosinophil count increased (Investigations) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Eye contusion (Injury, poisoning and procedural complications) | 0 | 1
Flushing (Vascular disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 0
Gastric pH decreased (Investigations) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 1
Hot flush (Vascular disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Illness (General disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 0
Injection site pain (General disorders) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1
Malaise (General disorders) | 0 | 1
Mean cell haemoglobin increased (Investigations) | 0 | 1
Mean cell volume increased (Investigations) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Protein urine (Investigations) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Temperature regulation disorder (General disorders) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary tract inflammation (Renal and urinary disorders) | 0 | 1
Urine flow decreased (Renal and urinary disorders) | 1 | 0
Weight increased (Investigations) | 0 | 1
White blood cell count increased (Investigations) | 0 | 1
Neutrophil count increased (Investigations) | 0 | 1
Renal cyst (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/52/NCT03750552/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-19): https://cdn.clinicaltrials.gov/large-docs/52/NCT03750552/SAP_001.pdf